CLINICAL TRIAL: NCT02381860
Title: Investigate the Effect of Tart Montmorency Cherry Juice (Prunus Cerasus) on Cerebral Blood Flow and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glyn Howatson, Dr, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NUKK2
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The PLA supplement consisted of a commercially available, less than 5% fruit, cordial (Protein - Trace, Carbohydrate 260 mg•mL-1, Sodium 0.02 mg•mL-1, Fibre-Trace and Anthocyanins-Trace for colour), mixed with water, whey protein isolate (Arla Foods Ltd., Leeds, UK) and maltodextrin (MyProtein Ltd., Northwich, UK) until matched for carbohydrate and calorie content of the MC.
  Interventions: Other: Placebo
- 60mL of cherry concentrate with 100ml water (Active Comparator): One bolus of 60mL of tart Montmorency cherry (MC) juice mixed with 100mL of water. Independent analysis of MC (Atlas Biosciences, 2010) provided the following compositional data; Fat 0.028 mg•mL-1, Protein 31.47 mg•mL-1, Carbohydrate 669.4 mg•mL-1, Cholesterol < 0.01 mg•mL-1, Sodium 0.691 mg•mL-1, Calcium 0.137 mg•mL-1 and Iron 0.026 mg•mL-1. Additionally, according to the manufacturers guidelines (Cherry Active, Hanworth, UK),
  Interventions: Dietary Supplement: 60mL tart Montmorency cherry juice

INTERVENTIONS:
Other: Placebo — One bolus of less than 5% fruit cordial mixed with water, maltodextrin and whey protein isolate to match for carbohydrate and calorie content of the juice.
  Other Names: less than 5% "Kia Ora" mixed fruit squash
  Arms: Placebo
Dietary Supplement: 60mL tart Montmorency cherry juice — One bolus of 60mL of tart Montmorency concentrate mixed with 100mL of water.
  Arms: 60mL of cherry concentrate with 100ml water

SUMMARY:
Scientific studies in humans suggest that diets high in fruit and vegetables may be able to improve some aspects of mental performance such as improving memory and reaction times. One reason that that these improvements may occur is that these compounds contain phytochemicals which may increase blood flow and, therefore, the delivery of oxygen and nutrients to the brain. If this is the case it is possible to measure this increased blood flow by a non-invasive technique called Near Infrared Spectroscopy. The purpose of this study is to examine the effect of a fruit juice on cerebral blood flow and cognitive function

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on three occasions. The first of these will be an initial screening/training visit, within 14 days of the first active study visit. During the initial visit participants will be provided with written informed consent and screened with regards the study exclusion/inclusion criteria. Training will be given on the cognitive tasks and familiarisation with the study procedures will be provided.

Study days: Forty - eight hours prior to each study day, participants will begin dietary restrictions. Participants will then attend the first study day following an overnight fast. A cannula will be inserted and baseline blood samples obtained, baseline measures of cerebral blood flow will be examined using near infrared spectroscopy and its effect on cognitive function using a cognitive demand battery. The relevant drink will then be provided and blood samples and blood flow measures will be taken at hourly intervals (1, 2, 3, and 5h). No additional food or drink will be provided during the study period except for low-nitrate mineral water. After a minimum of 2 weeks, participants will be asked to return to the lab and repeat the procedure with the other drink.

Cerebrovascular Responses

Cerebral oxygenation will be assessed using near - infrared spectroscopy . Two near-infrared sensors will be placed on the skin over the right and left prefrontal cortex region of the forehead, and the signals were averaged to determine cerebral oxygenation. The sensors will be secured to the skin using double-sided adhesive tape and shielded from ambient light using an elastic bandage. The sensors alternately emit near-infrared light at wavelengths of 730 and 810 nm. Each sensor contains two detectors located at 3 and 4 cm from the emitting source that detect oxygenated and deoxygenated states of Hb to estimate regional O2 saturation based on internal algorithms (Rasmussen et al. 2007).

Blood velocity in the middle cerebral artery (MCAV) will be determined using transcranial Doppler sonography. A 2 MHz Doppler probe was positioned over the right middle cerebral artery using previously described search techniques (Aaslid et al. 1982) and will be secured with an adjustable headset (DiaMon, Compumedics DWL). The mean depth for Doppler signals was 51 ± 3 mm. Arterial blood pressure will be recorded with a transducer located at heart level (TruWave, Edwards Lifesciences, Nyon, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40-60 years
* Not currently taking any medication

Exclusion Criteria:

* Those aged <40 or >60 years
* Currently taking medication

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in Cerebral Blood Flow | 0,1,2,3, and 5 hours

SECONDARY OUTCOMES:
Changes in Cognitive Function | 0,1,2,3 and 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle, United Kingdom